CLINICAL TRIAL: NCT03780088
Title: Improving Access to Care: Testing an Integrated Care Mobile Health Intervention to Improve Sleep and Mental Health in Adolescents
Brief Title: Improving Access to Care: Testing an Integrated Care Mobile Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46142
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Insomnia; Delayed Sleep Phase
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mTranS-C (Experimental): Access to a mobile and computer accessible adaptation of Transdiagnostic Sleep and Circadian Intervention
  Interventions: Behavioral: mTranS-C

INTERVENTIONS:
Behavioral: mTranS-C — mobile health

SUMMARY:
This study aims to evaluate the feasibility, effectiveness, and dissemination potential of an innovative strategy for improving access to effective sleep health care for adolescents. The study will test an adaptation of the Transdiagnostic Sleep and Circadian Intervention (TranS-C), a brief sleep intervention with demonstrated efficacy for improving sleep and mental health outcomes in youth.

DETAILED DESCRIPTION:
This adaptation is designed to address the following key challenges to accessing care: (1) to overcome the challenge of low availability of qualified providers as a barrier to treatment access, we have adapted TranS-C for online and mobile device delivery (referred to as mTranS-C), thereby leveraging the high rates of mobile phone and internet use in adolescents; (2) to further increase access we will disseminate mTranS-C within primary care services, a proven strategy for improving access to behavioral health care; and (3) we focus on low-income communities, where there is a higher prevalence of sleep problems and low access to services.

ELIGIBILITY:
Inclusion Criteria:

* age 12-18 years
* a sleep health deficit
* youth has access to a mobile phone or internet
* youth is fluent in English.

Exclusion Criteria:

* current use of medications or herbs with known effects on sleep
* current substance use disorder
* current suicidality/thoughts of death
* thought disorder
* unstable major medical conditions
* current psychotherapy for sleep health deficits

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | baseline to end of treatment (anticipated average exposure 2 months), and month 5
  A validated questionnaire; total score range between 0 and 21, with higher numbers representing worse sleep quality.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | baseline to end of treatment (anticipated average exposure 2 months), and month 5
  A validated questionnaire measuring depressive symptom severity. The total score ranges between 0 and 19. Scores are rated as minimal (0-4), mild (5-9), moderate (10-14), and severe (15-19).
Strengths & Difficulties Questionnaire (SDQ) | baseline and at months 2 and 5
  The Strengths and Difficulties Questionnaire (SDQ) is a validated 25 item behavioral screening questionnaire. Individual items are rated 'Somewhat True' (always scored as 1), 'Not True'(score is typically 0 except when reverse scored) and 'Certainly True' (score is typically 2 except when reverse scored). The SDQ comprise 5 scales (Prosocial, Peer Problems, Hyperactivity, Conduct and Emotional Problems) of 5 items each. For each of the 5 scales the score can range from 0 to 10 if all items were completed. These scores can be scaled up pro-rata if at least 3 items were completed, e.g. a score of 4 based on 3 completed items can be scaled up to a score of 7 (6.67 rounded up) for 5 items. A total difficulties score is generated by summing scores from all the scales except the prosocial scale. The resultant score ranges from 0 to 40, and is counted as missing of one of the 4 component scores is missing.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Asarnow, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Gardner Packard Children's Health Center, Atherton, California, United States

IPD SHARING:
Plan to Share IPD: No